CLINICAL TRIAL: NCT01408329
Title: Effects of Cyclic Variations in Altitude Conditioning (CVAC) on Wellness and Activity Measures
Acronym: CVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Anne Friedlander, Consulting Professor, Palo Alto Veterans Institute for Research
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FRI0016
Record Dates: First submitted 2011-07-28; First posted 2011-08-03 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-08

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Sham altitude changes - The CVAC device consists of a small pod-like chamber attached to a computer system that controls a strong pump that can draw air rapidly out of the chamber to increase the simulated altitude. The sham-treated group (SH) was exposed to regular, slowly-fluctuating pressures that reached a maximum altitude of 607 m for all 30 sessions. Sham sessions mimicked the noises and initial pressure-change sensations created in the active sessions, thus giving naıve subjects the impression that they were experiencing altitude treatment. All subjects were blind to their elevation throughout the intervention.
  Interventions: Device: CVAC Device (Cyclic Variations in Altitude Conditioning)
- Hypoxic intervention (Experimental): Cyclic Hypobaric Hypoxia (CHH) subjects were given 40 min sessions inside the CVAC device per day (two 20 min sessions sequentially per day), 3 days a week for 10 weeks, for a total of 30 sessions or 20 hours. After familiarization sessions, pre-programmed sessions were administered, progressing from Tier 1 to 5. Subjects rotated through three pre-programmed sessions per Tier and each session varied the pattern and rate of hypoxic fluctuations, so that subjects would experience a constantly changing stimulus at each elevation. Five weeks were allotted to progress from Tier 1 (3048 m) to Tier 4 (5486 m). At Tier 5 (6096 m), there was an additional 5 weeks of exposure.
  Interventions: Device: CVAC Device (Cyclic Variations in Altitude Conditioning)

INTERVENTIONS:
Device: CVAC Device (Cyclic Variations in Altitude Conditioning) — A hypobaric hypoxia chamber

SUMMARY:
Cyclic Variation in Altitude Conditioning (CVAC) is a new technique that uses a pod-like device to expose users to controlled fluctuations in air pressure. It is designed to promote quicker altitude acclimatization, thus promoting improvements in exercise capacity at altitude and, possibly, at sea level. However, over the past few years, anecdotal stories from users of the device suggest that the CVAC treatments might be causing changes beyond the expected endurance exercise performance benefits. Therefore, the purpose of the study is to obtain data on some of the previous anecdotal claims regarding the device (e.g. increases in strength, improved glucose tolerance, reduction of neuropathic pain and decreased joint swelling) as well as to obtain broad questionnaire data in order to identify more specific variables to investigate in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy middle aged men at risk for metabolic syndrome

Exclusion Criteria:

* Uncontrolled hypertension,
* sensitive ears,
* anything that would preclude person from sustaining rapid pressure changes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Friedlander, PhD, Principal Investigator — Veterans Affairs Palo Alto Health Care System

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Palo Alto and surrounding areas by flyer and advertisement
Pre-assignment Details: Medical Screening Group Matching by 3rd party
Groups:
- Sham Group: Slowly fluctuating pressures simulating altitude up to 607 meters
- Cyclic Hypoxic Group: Rapidly fluctuating pressures simulating altitude up to 6096 meters
Period: Overall Study
Arm/Group | Sham Group | Cyclic Hypoxic Group
Started | 13 | 15
Completed | 10 | 11
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Group | Cyclic Hypoxic Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (4) | 48 (6) | 49 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose Concentration
Time Frame: Glucose measurements were made at baseline, 3, 6, & 10 weeks. Blood was collected consistently after a 10-12 h fast the morning after a CVAC session (except for baseline).
Population: Those that completed the study
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Cyclic Hypoxic Group: Rapidly fluctuating pressures simulating altitude up to 6097m
Arm/Group | Sham Group | Cyclic Hypoxic Group
Number analyzed (Participants) | 10 | 11
mg/dl
  Baseline | 93.8 (7.6) | 95.7 (9.0)
  3 weeks | 94.1 (6.2) | 93.3 (8.5)
  6 weeks | 95.3 (7.5) | 92.5 (4.3)
  10 weeks | 96.8 (8.9) | 90.8 (6.9)

ADVERSE EVENTS:
Time Frame: The events occured over the 1 year period of the study
Description: The events did not require medical attention, but prevented the subjects from advancing to the higher levels of altitude exposure
Groups:
- Sham Group: Slowly fluctuating simulated altitude up to 607 meters.
- Cyclic Hypoxic Group: Rapidly fluctuating simulated altitude up to 6097 meters
Arm/Group | Sham Group | Cyclic Hypoxic Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Group (N=13) | Cyclic Hypoxic Group (N=15)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 3 (3) — 3 subjects felt ear pain with the changing pressure caused by the cyclic hypoxia and did not wish to continue to the highest elevation tiers.

LIMITATIONS AND CAVEATS:
Small Sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No